CLINICAL TRIAL: NCT00006187
Title: The Safety and Efficacy of an Investigational Drug in Delaying the Progression of Alzheimer's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0025
Record Dates: First submitted 2000-08-25; First posted 2000-08-28 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2003-10

CONDITIONS: Alzheimer Disease
Keywords: Investigational Drug
MeSH Terms: conditions — Alzheimer Disease | interventions — Drugs, Investigational

INTERVENTIONS:
Drug: Investigational drug

SUMMARY:
This is a 15-month study with two phases. During the first 12-month phase of this study, patients will be randomly assigned to receive either active study drug or placebo (approximately half of all patients will be on active study drug, the other half on placebo). The second phase is a 3-month randomized withdrawal period. For this phase approximately 10% of the patients will remain on the active drug.

DETAILED DESCRIPTION:
This is a placebo-controlled, parallel-groups, 12 month, double-blind study, followed by a 3-month, double-blind, randomized withdrawal period to evaluate the efficacy and safety of an investigational drug (currently approved for other indications) to slow the progression of symptoms of AD. Patients with probable AD according to NINCDS-ADRDA criteria who have a Mini Mental State Examination (MMSE) score between 13 and 26 inclusive will be eligible for participation in the study.

Patients on stable doses of marketed cholinesterase inhibitors approved for the treatment of AD (except for tacrine) for at least 3 months are eligible for study entry. Use of NSAIDs (except aspirin 81 mg per day) is not allowed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female and at least 50 years of age or older
* Female patients must be postmenopausal or surgically sterilized
* Clinical diagnosis of AD
* Patient must be in good health except for AD diagnosis
* Patient must have informant/caregiver who can monitor and assist patient during the study

Exclusion Criteria:

* Patient is living in a nursing home or skilled nursing facility
* Women will be ineligible if not postmenopausal or surgically sterilized
* Site physician or Sponsor may exclude patients with serious medical problems such as cancer, cardiovascular disease, major neurological or psychiatric illness, thyroid disease, or major head trauma

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2005-06 (Estimated); Study Completion 2005-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Beck, MD, PhD, Principal Investigator — Merck Sharp & Dohme LLC
Locations (34):
- United States (34):
  - Pivotal Research Centers, Peoria, Arizona
  - California Clinical Trials, Beverly Hills, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Daniel Grosz MD, Northridge, California
  - Pharmacology Research Institute, Riverside, California
  - Pacific Research Network, San Diego, California
  - San Francisco Headache Clinic, San Francisco, California
  - Yale University, Alzheimer's Disease ResearchUnit, New Haven, Connecticut
  - New England Center for Headache, Stamford, Connecticut
  - Baumel-Eisner Neuromedical Institute, Boca Raton, Florida
  - Baumel-Eisner Neuromedical Institute, Fort Lauderdale, Florida
  - ICSL Clinical Studies, Fort Myers, Florida
  - ICSL Clinical Studies, Melbourne, Florida
  - ICSL Clinical Studies, Sarasota, Florida
  - ICSL Clinical Studies, St. Petersburg, Florida
  - Meridien Research, St. Petersburg, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Palm Beach Neurological Center, West Palm Beach, Florida
  - Chicago Center for Clinical Research, Chicago, Illinois
  - ICSL Clinical Studies, South Yarmouth, Massachusetts
  - Las Vegas Center for Clinical Research, Las Vegas, Nevada
  - Nathan Klein Institute, Orangeburg, New York
  - University of Rochester, Rochester, New York
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Pahl Brain Associates, P.C., Oklahoma City, Oklahoma
  - Clinical Pharmaceutical Trials, Tulsa, Oklahoma
  - Pacific NW Clinical Research Center, Portland, Oregon
  - Institute for Advanced Clinical Research, Elkins Park, Pennsylvania
  - ICSL Clinical Studies, Philadelphia, Pennsylvania
  - ICSL Clinical Studies, East Providence, Rhode Island
  - Pharmacology Research Clinic, Salt Lake City, Utah
  - Seattle Clinical Research Center, Seattle, Washington
  - Froedtert Lutheran Memorial Hospital, Milwaukee, Wisconsin